CLINICAL TRIAL: NCT04095078
Title: Efficiency and Acceptability of SIMEOX® Used Autonomously at Home for Bronchial Clearance in Patients With Cystic Fibrosis: Ancillary Study
Brief Title: Ancillary Home Airway Clearance in CF Patients ( HomeCareSIMEOX )
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physio-Assist (Industry)
Collaborators: Icadom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ancillary Home-Care SIMEOX
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Pulmonary Cystic Fibrosis
Keywords: bronchial clearance; cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, multicenter trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIMEOX (Experimental): Use the device for 3 months in addition to usual care
  Interventions: Device: SIMEOX
- Control (No Intervention): Usual care

INTERVENTIONS:
Device: SIMEOX — Use without obligation, in autonomous and at home of the bronchial clearance device: SIMEOX
  Arms: SIMEOX

SUMMARY:
Regular bronchial clearance is essential in patients with cystic fibrosis for their bronchial health. SIMEOX® (Physio-Assist, Aix en Provence, France) is an innovative medical device for the drainage of the bronchial tree. By changing the rheological properties of mucus, SIMEOX® helps to mobilize secretions and assists their transport to the upper airways. This technology is based on fundamental research on bronchial mucus rheology. At the present time, SIMEOX® device is mainly used over a short period at the time or after an exacerbation in healthcare structures (hospitals, physiotherapy practices, postcare, and rehabilitation units, etc…). The clinical effects observed in the short term encourages long-term autonomous use by the patients themselves. The overall objective of this study is to evaluate the efficiency and acceptability of SIMEOX® used at home by the patient himself for bronchial clearance in patients with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* one of the 56 first patients of HOME-CARE SIMEOX study
* same criteria as HOME-CARE SIMEOX study

Exclusion Criteria:

* same criteria as HOME-CARE SIMEOX study

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Pulmonary static hyperinflation assessed by residual volume | Change from baseline at 3 months
  Relative variation in Pulmonary residual volume in the SIMEOX® treated group versus control group.

SECONDARY OUTCOMES:
Use assessed by the duration of use of SIMEOX® device | During 3 months of use
  Assess the duration of uses of the device SIMEOX by the patient in the SIMEOX® treated group to assess the use by patient of the device.
Inspiratory capacity | Change from baseline at 3 months
  Relative variation of Inspiratory capacity in liter in the SIMEOX® treated group versus control group
Residual functional capacity (RFC) | Change from baseline at 3 months
  Relative variation of Residual functional capacity (RFC) in liter in the SIMEOX® treated group versus control group
Total lung capacity (TLC) | Change from baseline at 3 months
  Relative variation of Total lung capacity (TLC) in liter in the SIMEOX® treated group versus control group

CONTACTS AND LOCATIONS:
Overall Officials: Boubou Camara, MD, Principal Investigator — CHUGA
Locations (5):
- France (5):
  - Grenoble University Hospital : pneumo-pediatric department, Grenoble
  - Grenoble University-Affiliated Hospital : Pneumology department, Grenoble
  - Montpellier Hospital Center, Montpellier
  - Nice University-Affiliated Hospital : Pneumology department, Nice
  - Nice University-Affiliated Hospital : Pneumo-pediatric department, Nice

IPD SHARING:
Plan to Share IPD: No